CLINICAL TRIAL: NCT00509067
Title: Interventions to Test the Alpha7 Nicotinic Receptor Model in Schizophrenia
Brief Title: Use of Galantamine and CDP-choline (Citicoline) to Treat Adults With Schizophrenia
Acronym: STAR-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Stephen I. Deutsch, Professor and Chair, Dept. of Psychiatry & Behavioral Sciences, Eastern Virginia Medical School, National Institute of Mental Health (NIMH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R34MH077849 (NIH); R34MH077849 (NIH); DATR A5-ETBD
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Results first posted 2014-02-07 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-02

CONDITIONS: Schizophrenia
Keywords: Schizoaffective Disorder; Acetylcholine; Nicotinic Receptors; Nicotine; Galantamine; negative symptoms
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Galantamine; Cytidine Diphosphate Choline; Risperidone; Olanzapine; Quetiapine Fumarate; ziprasidone; Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Participants assigned to receive galantamine and CDP-choline
  Interventions: Drug: Galantamine; Drug: CDP-choline; Drug: risperidone, olanzapine, quetiapine, ziprasidone, and/or aripiprazole
- B (Placebo Comparator): Participants assigned to receive placebo
  Interventions: Drug: Placebo; Drug: risperidone, olanzapine, quetiapine, ziprasidone, and/or aripiprazole

INTERVENTIONS:
Drug: Galantamine — Galantamine will be titrated to 24 mg/day over 2 weeks. Participants will receive 8 mg/day in two divided doses for 1 week, 16 mg/day in two divided doses for 1 week, and 24 mg/day in two divided doses beginning in Week 3. They will be maintained on 24 mg/day for the remainder of the study.
  Other Names: Razadyne
  Arms: A
Drug: CDP-choline — CDP-choline will serve as the dietary source of choline. CDP-choline will be titrated to 2000 mg/day over 1 week. Subjects will receive 500 mg/day for 3 days; Thereafter, the dose of CDP-choline will be increased to 1,000 mg/day in two divided doses for 4 days. At the beginning of Week 2, participants will receive the maximum fixed dose of 2000 mg/day in two divided doses, which will be held constant through the end of Week 16.
  Arms: A
Drug: Placebo — The schedule of dose titration of placebo galantamine and placebo CDP-choline will follow the schedule of active medication condition using matching placebos for each agent.
  Arms: B
Drug: risperidone, olanzapine, quetiapine, ziprasidone, and/or aripiprazole — All participants will continue to take their regular regimen of risperidone, olanzapine, quetiapine, ziprasidone, and/or aripiprazole throughout the trial in addition to their assigned treatment.

SUMMARY:
This study will evaluate the effectiveness of galantamine and CDP-choline in improving symptoms associated with schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a life-long brain disorder affecting approximately 1 percent of Americans each year. Schizophrenia can be extremely disabling, causing people to hear voices, experience paranoia or hallucinations, believe that others are controlling their thoughts, and even fail at maintaining a job or caring for themselves. Current medications help to relieve most of these negative symptoms, but not all. Many people with schizophrenia still suffer from low energy levels, an inability to concentrate, and memory loss. Galantamine is a medication that is used to improve memory and energy levels in people with Alzheimer's disease, and CDP-choline is a nutritional supplement. The purpose of this study is to evaluate the effectiveness of adding galantamine and CDP-choline to a stable anti-psychotic medication regimen of risperidone as a way of improving symptoms in adults with schizophrenia.

Participants in this double-blind study will attend an initial screening during which they will undergo a physical exam, an electrocardiogram, and blood and urine collection. Participants will then be randomly assigned to receive galantamine and CDP-choline or a placebo treatment for 16 weeks. Participants assigned to the treatment group will take 500 mg of CDP-choline daily for the first 3 days, 1,000 mg daily for the next 4 days, and 2,000 mg daily for the following 15 weeks. Participants assigned to the treatment group will also take 8 mg of galantamine daily for the first week, 16 mg daily for the next week, and 24 mg daily for the following 14 weeks. Participants assigned to the control group will take two types of placebo pills every day for 16 weeks. All participants will continue to take their regular regimen of risperidone, olanzapine, quetiapine, ziprasidone, and/or aripiprazole throughout the trial in addition to their assigned treatment. Staff members will meet with participants during the first week of the study and every 4 weeks afterward until study completion. During these meetings, participants will identify any side effects, report nicotine intake, breathe into a machine that measures the amount of nicotine in the body, and complete written and computerized tasks on concentration and memory. Each meeting may last up to 3 hours. On the last week of the study, blood and urine samples will be collected and an electrocardiogram will be administered. Results from this study will be used to evaluate whether CDP-choline and galantamine improve schizophrenia symptoms.

CDP-choline and matching placebos were purchased from LifeLink Corporation. Galantamine and matching placebos were prepared and donated by Ortho McNeil Janssen Scientific Affairs LLC.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for schizophrenia or schizoaffective disorder
* Eligible for care within the Veterans Affairs Medical system
* Taking risperidone, olanzapine, quetiapine, ziprasidone, and/or aripiprazole (oral or injection)

Exclusion Criteria:

* Significant liver, kidney, lung, endocrine, active peptic ulcer, or cardiovascular disease
* Seizure disorder and/or head injury
* Substance use or abuse within 3 months of study entry
* Pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2007-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen I. Deutsch, PhD, MD, Principal Investigator — Washington Veterans Affairs Medical Center
Locations (1):
- Washington Veterans Affairs Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Deutsch SI, Schwartz BL, Schooler NR, Rosse RB, Mastropaolo J, Gaskins B. First administration of cytidine diphosphocholine and galantamine in schizophrenia: a sustained alpha7 nicotinic agonist strategy. Clin Neuropharmacol. 2008 Jan-Feb;31(1):34-9. doi: 10.1097/wnf.0b013e31806462ba. PMID 18303489
- [Background] Deutsch SI, Rosse RB, Schwartz BL, Schooler NR, Gaskins BL, Long KD, Mastropaolo J. Effects of CDP-choline and the combination of CDP-choline and galantamine differ in an animal model of schizophrenia: development of a selective alpha7 nicotinic acetylcholine receptor agonist strategy. Eur Neuropsychopharmacol. 2008 Feb;18(2):147-51. doi: 10.1016/j.euroneuro.2007.05.008. Epub 2007 Jul 26. PMID 17656074
- [Background] Martin LF, Freedman R. Schizophrenia and the alpha7 nicotinic acetylcholine receptor. Int Rev Neurobiol. 2007;78:225-46. doi: 10.1016/S0074-7742(06)78008-4. PMID 17349863
- [Background] Olincy A, Harris JG, Johnson LL, Pender V, Kongs S, Allensworth D, Ellis J, Zerbe GO, Leonard S, Stevens KE, Stevens JO, Martin L, Adler LE, Soti F, Kem WR, Freedman R. Proof-of-concept trial of an alpha7 nicotinic agonist in schizophrenia. Arch Gen Psychiatry. 2006 Jun;63(6):630-8. doi: 10.1001/archpsyc.63.6.630. PMID 16754836
- See also: Link for publication of study results — http://dx.doi.org/10.1016/j.schres.2013.05.023

RESULTS

PARTICIPANT FLOW:
Groups:
- Galantamine/CDP Choline: Participants assigned to receive galantamine and CDP-choline
- Placebos for Galantamine/CDP Choline: Participants assigned to receive placebo
Period: Overall Study
Arm/Group | Galantamine/CDP Choline | Placebos for Galantamine/CDP Choline
Started | 19 | 24
Completed | 15 | 19
Not Completed | 4 | 5
Not completed — Lost to Follow-up | 1 | 1
Not completed — Adverse Event | 3 | 1
Not completed — Protocol Violation | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Galantamine/CDP Choline | Placebos for Galantamine/CDP Choline | Total
Number analyzed (Participants) | 19 | 24 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 22 | 41
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.37 (8.50) | 52.38 (11.04) | 53.28 (9.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 17 | 22 | 39
Region of Enrollment [Number; unit: participants]
  United States | 19 | 24 | 43

OUTCOME MEASURES:

1. Primary Outcome: Negative Symptoms Measured on Positive and Negative Syndrome Scale (PANSS)
Description: The score for each subject was the sum of the ratings for five items on the negative-symptom subscale of the PANSS: 1) blunted affect, 2) emotional withdrawal, 3) poor rapport, 4) passive/apathetic social withdrawal, and 5) lack of spontaneity and flow of conversation. Each item (symptom) is rated on a scale from 1 = absence of negative symptom to 7 = extreme negative symptom. The sum of the ratings for the five items range from 5 to 35, with higher scores indicating more severe symptoms. The primary outcome measure is the mean of the sum of these ratings across subjects.
Time Frame: Measured at Baseline and Weeks 4, 8, 12, and 16
Population: intent to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Galantamine/CDP Choline | Placebos for Galantamine/CDP Choline
Number analyzed (Participants) | 19 | 24
units on a scale
  Baseline | 17.63 (3.48) | 18.29 (4.52)
  Week 4 | 17.06 (5.6) | 17.08 (5.64)
  Week 8 | 13.93 (5.09) | 17.26 (5.8)
  Week 12 | 14.93 (5.2) | 17.32 (5.21)
  Week 16 | 13.93 (5.2) | 16.05 (5.97)

2. Secondary Outcome: Clinical Global Impression
Description: The score for each subject was the mean rating on the severity item. The score of the item ranged from 1 (normal) to 7 (among most severely ill).
Time Frame: Measured at Baseline and Weeks 4, 8, 12, and 16
Population: intent to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Galantamine and CDP-choline Group: Participants assigned to galantamine and CDP-choline
  Galantamine: Galantamine will be titrated to 24 mg/day over 2 weeks. Participants will receive 8 mg/day in two divided doses for 1 week, 16 mg/day in two divided doses for 1 week, and 24 mg/day in two divided doses beginning in Week 3. They will be maintained on 24 mg/day for the remainder of the study.
  CDP-choline: CDP-choline will serve as the dietary source of choline. CDP-choline will be titrated to 2000 mg/day over 1 week. Subjects will receive 500 mg/day for 3 days; Thereafter, the dose of CDP-choline will be increased to 1,000 mg/day in two divided doses for 4 days. At the beginning of Week 2, participants will receive the maximum fixed dose of 2000 mg/day in two divided doses, which will be held constant through the end of Week 16.
  risperidone, olanzapine, quetiapine, ziprasidone, and/or aripiprazole: All participants will continue to take their regular regimen of risperidone, olanzapine, quetiapine, zipr
- Placebo Group: Participants assigned to placebo
  Placebo: The schedule of dose titration of placebo galantamine and placebo CDP-choline will follow the schedule of active medication condition using matching placebos for each agent.
  risperidone, olanzapine, quetiapine, ziprasidone, and/or aripiprazole: All participants will continue to take their regular regimen of risperidone, olanzapine, quetiapine, ziprasidone, and/or aripiprazole throughout the trial in addition to their assigned treatment.
Arm/Group | Galantamine and CDP-choline Group | Placebo Group
Number analyzed (Participants) | 19 | 24
units on a scale
  Baseline | 4.32 (.48) | 4.38 (.58)
  Week 4 | 4 (.49) | 3.92 (.65)
  Week 8 | 3.67 (.62) | 4.04 (.82)
  Week 12 | 3.87 (.64) | 4 (.82)
  Week 16 | 3.8 (.68) | 3.68 (.67)
Statistical Analysis 1: Comparison: Galantamine and CDP-choline Group vs Placebo Group; Test type: Superiority; p = 0.93, Mixed Models Analysis — alpha set at P < .05; Time (0, 4, 8, 12, 16 wks) x Treatment (Drug, Placebo) Effect: F(1, 33)=0.01

3. Secondary Outcome: MATRICS Verbal Learning and Memory
Description: The measure of verbal learning and memory is the Hopkins Verbal Learning Test. The score for each subject is the sum of the total number of words recalled correctly for Trials 1, 2, and 3. The measure is the mean of these scores at baseline, Week 8, and Week 16.
Time Frame: Measured at Baseline and Weeks 8 and 16
Population: intent to treat
Measure: Mean (Standard Deviation); unit: raw scores
Groups:
- Galantamine and CDP-choline Group: Participants assigned to receive galantamine/CDP-choline
  Galantamine: Galantamine will be titrated to 24 mg/day over 2 weeks. Participants will receive 8 mg/day in two divided doses for 1 week, 16 mg/day in two divided doses for 1 week, and 24 mg/day in two divided doses beginning in Week 3. They will be maintained on 24 mg/day for the remainder of the study.
  CDP-choline: CDP-choline will serve as the dietary source of choline. CDP-choline will be titrated to 2000 mg/day over 1 week. Subjects will receive 500 mg/day for 3 days; Thereafter, the dose of CDP-choline will be increased to 1,000 mg/day in two divided doses for 4 days. At the beginning of Week 2, participants will receive the maximum fixed dose of 2000 mg/day in two divided doses, which will be held constant through the end of Week 16.
  risperidone, olanzapine, quetiapine, ziprasidone, and/or aripiprazole: All participants will continue to take their regular regimen of risperidone, olanzapine, quetiapine, zipr
- Placebo Group: Participants assigned to receive placebo
  Placebo: The schedule of dose titration of placebo galantamine and placebo CDP-choline will follow the schedule of active medication condition using matching placebos for each agent.
  risperidone, olanzapine, quetiapine, ziprasidone, and/or aripiprazole: All participants will continue to take their regular regimen of risperidone, olanzapine, quetiapine, ziprasidone, and/or aripiprazole throughout the trial in addition to their assigned treatment.
Arm/Group | Galantamine and CDP-choline Group | Placebo Group
Number analyzed (Participants) | 19 | 24
raw scores
  Baseline | 20.5 (5.1) | 20.6 (5.8)
  Week 8 | 21.8 (4.6) | 21.2 (5.9)
  Week 16 | 23.0 (4.7) | 20.4 (5.4)
Statistical Analysis 1: Comparison: Galantamine and CDP-choline Group vs Placebo Group; Test type: Superiority; p = 0.23, Mixed Models Analysis — alpha level set at .05; Time (0, 8, 16 weeks) x Group (Drug, Placebo) Effect: F(1, 32.8)=1.48
Statistical Analysis 2: Comparison: Galantamine and CDP-choline Group vs Placebo Group; Test type: Superiority; p = 0.23, Mixed Models Analysis — alpha set at P<0.05; Time (0, 8, 16, weeks) x Group (Drug, Placebo) Effect: F(1, 32.8)=1.48

ADVERSE EVENTS:
Time Frame: Adverse events were collected weekly over 16 weeks for each participant.
Description: Table presents adverse events by group that were at least moderate at any time point.
  All AEs were assessed (systematic assessment) on a scale from 1 = absent to 4 = severe.
Arm/Group | Galantamine/CDP Choline | Placebos for Galantamine/CDP Choline
Serious Adverse Events (participants affected / at risk) | 0/19 | 1/24
Other Adverse Events (participants affected / at risk) | 10/19 | 14/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galantamine/CDP Choline (N=19) | Placebos for Galantamine/CDP Choline (N=24)
hospitalized for cardiac symptoms (Cardiac disorders) | 0 (0) | 1 (1) — One placebo participant was hospitalized with cardiac symptoms. This SAE resolved.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Galantamine/CDP Choline (N=19) | Placebos for Galantamine/CDP Choline (N=24)
Abdominal Pain (Gastrointestinal disorders) | 6 | 3
Drowsiness (General disorders) | 6 | 3
Headache (General disorders) | 5 | 5
Malaise (General disorders) | 5 | 2
Restlessness (General disorders) | 5 | 2
Dry Mouth (General disorders) | 4 | 4
Indigestion (Gastrointestinal disorders) | 4 | 1
Nausea (Gastrointestinal disorders) | 4 | 3
Sleep problem (General disorders) | 4 | 3
Excess Salivation (General disorders) | 3 | 4
Insomnia (General disorders) | 3 | 2
Nasal Congestion (General disorders) | 3 | 4
Sweating (General disorders) | 3 | 5
Syncope (Cardiac disorders) | 3 | 2
Decrease in Appetite (Gastrointestinal disorders) | 2 | 2
Diarrhea (Gastrointestinal disorders) | 2 | 4
Fever (General disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes